CLINICAL TRIAL: NCT06560463
Title: Comparison of Continous Glucose Monitor and OGTT as a Screen for Cystic Fibrosis Related Diabetes and Impaired Glucose Tolerance
Brief Title: Continuous Glucose Monitoring and OGTT Screen for Cystic Fibrosis Related Diabetes in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Julie Biller, Chief, Professor | Medicine, Medical College of Wisconsin
Other Study IDs: PRO00051083
Record Dates: First submitted 2024-07-02; First posted 2024-08-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cystic Fibrosis
  Interventions: Device: Access to Dexcom G7 CGM Data

INTERVENTIONS:
Device: Access to Dexcom G7 CGM Data — Eligible patients will undergo Continuous Glucose Monitoring using the Dexcom G7

SUMMARY:
Cystic Fibrosis (CF) related diabetes (CFRD) is a unique form of diabetes mellitus, different from type 1 diabetes and type 2 diabetes. The diagnosis of CFRD is associated with a decline in pulmonary function, decreased nutritional status, and increased mortality. CFRD is extremely common in people with CF, occurring in approximately 40-50% of adults with CF. Impaired glucose tolerance or dysglycemia is also very common in CF. It is standard of care to screen for CFRD annually from the age of 10 years with a two-hour Oral Glucose Tolerance Test (OGTT) with 75 g dextrose. The gold standard screening for CFRD is the OGTT which is problematic as it is time consuming for patient and staff and adherence to annual screening is low among CF centers.

Survival has improved dramatically with the advent of CFTR modulators and it is presumed that the incidence of CFRD will increase with increased life expectancy. The Cystic Fibrosis Foundation (CFF) has developed the oldest disease specific patient registry, consisting of approximately 35000 patients, so there is vast historical information available on individual patients and larger datasets on the CF community as a whole. Based on the 2021 CFF patient registry data, the current life expectancy for CF patients born between 2017 and 2021 is 53 years - a 15 year increase from a decade ago.

DETAILED DESCRIPTION:
Research design and methods

* Clinic will continue to follow CFF standard of care guidelines. Subjects will complete the annual OGTT and an annual HgbA1c.
* Sample Dexcom G7 Sensors will be provided to the subjects for 10 day wear during a routine CF clinic appointment.
* The clinic RD will provide education on sensor application and assist the subjects in applying the sensors during the CF clinic visit.
* The clinic RD will assist subjects with install of phone applications (Dexcom G7 and Dexcom Clarity) to track data and produce reports. The interpretation of reports will be reviewed with the subjects.
* The clinic RD will review dietary sources of carbohydrates and request patients add notes with estimation of carbohydrate (g) intake in Dexcom G7 app for the 10 days
* The clinic RD will set up accounts for the subjects to share data in the Dexcom Clarity online platform.
* After 10 days of CGM wear the clinicians will review reports for time in range (TIR), incidence of hypoglycemia, % readings of hyperglycemia, glycemic variability.
* Clinic RD will also record subject body weight trajectory and if a CFTR modulator is prescribed.
* Data will be entered in RedCap for direct comparison of CGM data, HGbA1c and OGTT results.

Relevant CF standard of care data that will be entered into redcap:

1. CF genetic mutations
2. Pancreatic sufficiency status
3. BMI trends
4. Number of CF exacerbations and severity
5. FEV1 trends
6. Glycohemoglobin levels
7. Lipid levels
8. 2 hour hypoglycemia on CF standard OGTT
9. Blood pressure trends
10. Patient age Statistical Justification for number of subjects: The research team will be able to recruit a maximum of 30 patients for the study who will use Continual Glucose Monitoring (CGM) for the duration of the study period. Given about 40% of CF patients are expected to develop CFRD, there will be adequate variability in the data and adequate sample size to assess diagnostic test performance in this group.

Data Analysis: Descriptive statistics of patient sample characteristics will be performed with mean, standard deviation for continuous variables and counts, percentages for categorical variables. Several diagnosis and screening test performance measures such as sensitivity, specificity, receiver operating characteristic curves, area under the curve, positive predictive value, negative predictive value will be applied in the study. The oral glucose tolerance test (OGTT) will be used as the gold standard and compared against continuous glucose monitoring (CGM) (I.E. glucose level, time in range (TIR), etc ), and used to determine whether CGM effectively screens for Cystic Fibrosis Related Diabetes

ELIGIBILITY:
Inclusion Criteria:

1. An adult patient, diagnosed with CF, established with Froedtert Multidisciplinary CF Clinic.
2. Normal glucose tolerance or impaired glucose tolerance per OGTT completed in 2024.
3. At healthy baseline status at time of CGM wear and OGTT.

Exclusion Criteria:

1. Diagnosed with CFRD and treating with diabetogenic medications.
2. s/p transplant
3. pregnancy
4. failure to wear CGM for entirety of 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Cystic Fibrosis, age 18 years and older, who receive care in the Froedtert and MCW Adult Cystic Fibrosis program.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose measurement | 10 days
  Blood glucose levels will be continuously monitored over a ten-day period using a Dexcom G7 continuous glucose monitor (CGM)

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided